CLINICAL TRIAL: NCT06099691
Title: Investigating Outcomes That Matter and the Suitability of PROMs for Older People Living With Frailty
Brief Title: Outcomes That Matter and Questionnaires for Older People With Frailty
Status: Completed | Type: Observational
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Collaborators: University of Exeter (Other)
Responsible Party: Sponsor
Other Study IDs: 329896
Record Dates: First submitted 2023-10-17; First posted 2023-10-25 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Frailty
Keywords: Patient Reported Outcome Measures; Qualitative Research; Frailty; Health Priorities; Quality of Life
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults with frailty: Participants will be interviewed about what matters to them. They will then give their opinions on questionnaires that aim to measure what matters to them.
  Interventions: Behavioral: Qualitative Interviews

INTERVENTIONS:
Behavioral: Qualitative Interviews — Participants will take part in one 90-minute interview (or two 45-minute interviews if preferred). The interview will have two sections. The first section will include discussion of what matters to participants. The second section will introduce PROMs which may be pertinent to measuring what matters. The participants will be helped to reflect on their relevance and usefulness to them.

SUMMARY:
The goal of this qualitative study is to investigate what matters to older people living with frailty, and how this can be measured using questionnaires (Patient Reported Outcome Measures, or "PROMs").

The research questions are:

1. What outcomes matter to older adults living with frailty?
2. What are participants' perceptions of PROMs that could measure these outcomes?

Our estimated sample will be 15 older adults, approximately 5 people living with mild frailty, 5 living with moderate frailty and 5 living with severe frailty. Participants will take part in one 90-minute interview.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 65
* Indication of frailty in one of the following ways:

  * Clinical diagnosis of frailty
  * Assessment of at least "4" on the Clinical Frailty Scale by a healthcare professional
* Having mental capacity to consent to participate as defined under the Mental Capacity Act (2005). This will be assessed in the telephone conversation prior to the interview by a researcher who has received Mental Capacity training
* Available to be interviewed by face-to-face interview at the National Institute of Health Research (NIHR) Exeter Clinical Research Facility or as a home visit, or as an online meeting

Exclusion Criteria:

* Not able to participate in face-to-face interview or use video call technology
* Not assessed as frail
* Not able to express thoughts and opinions in sufficient depth for analysis, even with facilitation by a relative or carer. This will be assessed in the telephone conversation with the researcher prior to the interview.
* Lacking capacity to consent to participate as defined under the Mental Capacity Act (2005). An individual would be unable to participate if they cannot:

  * Understand the information relevant to the decision of participating
  * Retain that information
  * Use or weigh up that information as part of the process of deciding whether to participate
  * Communicate their decision to other people

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older people (aged 65 and over) living with frailty.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Identify outcomes that matter to older people with frailty | 6 months
  Qualitative interviews will be conducted with older people living with frailty to identify what matters to people (e.g. managing pain, functional independence, suitability of medications, social support). This may vary at different severities of frailty.
Investigate perceptions of questionnaires | 6 months
  Qualitative interviews will be conducted with older people living with frailty to investigate participants' perceptions of PROMs (questionnaires) that could measure outcomes that matter to them.

CONTACTS AND LOCATIONS:
Overall Officials: Suzy Hope, Principal Investigator — Royal Devon and Exeter NHS Foundation Trust
Locations (1):
- Royal Devon Hospital, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No